CLINICAL TRIAL: NCT04038112
Title: A Case Series of Method of Levels (MOL) Therapy for People Experiencing Psychosis
Brief Title: Method of Level (MOL) Therapy for Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jadwiga Nazimek, Clinical Psychology Trainee, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 257300
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: systematic case replication series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Method of Levels (MOL) (Other): all participants will be offered intervention
  Interventions: Other: psychological therapy Method of Levels (MOL)

INTERVENTIONS:
Other: psychological therapy Method of Levels (MOL) — Transdiagnostic, cognitive psychological therapy Method of Levels (MOL)

SUMMARY:
The study is a systematic case replication series of a new psychological therapy Method of Levels (MOL) for people who experience psychosis. Between 6 and 8 people with psychosis who receive services from CMHT will be recruited. Participants will complete baseline questionnaires measuring their symptoms and distress and will be offered up to 12 sessions of MOL. Following the completion of therapy they will complete the questionnaires measuring symptoms and distress again.

DETAILED DESCRIPTION:
Psychosis is an enduring and distressing mental illness which can cause high levels of disability. Recommended treatments include antipsychotic medication and Cognitive Behaviour Therapy (CBT). Antipsychotic drugs cause serious negative side effects which are intolerable for some patients. CBT can be difficult to conduct in the presence of comorbid problems and can be too demanding for some patients. Both medication and CBT sometimes fail to sufficiently reduce the symptoms. Method of Levels (MOL) is a flexible, short-term, cognitive therapy informed by a theory that explains the underpinnings of psychological distress and the mechanisms of action in effective therapy. The purpose of the current study is to evaluate the utility of MOL for individuals with non-affective psychosis who are under the care of secondary mental health services. A case series will explore the efficacy of MOL for the levels of symptoms, distress and general functioning. MOL will be offered to 6-8 individuals with psychosis within a flexible appointment scheduling system. Levels of symptoms, distress and general functioning will be measured before and after treatment. Open feedback interviews following the completion of treatment will allow us to evaluate the patients' experience of MOL. The project will provide preliminary data which will inform clinical practice and contribute to large scale research of MOL.

ELIGIBILITY:
Inclusion Criteria:

* Participants have to be registered with a Community Mental Health Services
* Participants need to either meet ICD-10 criteria for schizophrenia, schizoaffective disorder and delusional disorder or meet entry criteria for an Early Intervention for Psychosis service.

Exclusion Criteria:

* Known moderate to severe learning disability
* Known organic basis of symptoms
* Known lack of capacity to consent to participating in research
* Lack of fluency in English (since MOL therapy will be conducted in English and due to use of standardised assessment tools). This will be determined by the researcher.
* Acute inpatient status
* A primary diagnosis of a drug or alcohol dependency
* Concurrent psychological therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Community Assessment of Psychic Experiences (CAPE) | 12 weeks
  Self-administered questionnaire, measure of symptoms of psychosis and associated distress. Total scores range from 42 to 168 on both dimensions (symptoms and distress). Higher scores indicate higher frequency of symptoms and higher distress.
Reorganization of Conflict Scale (ROC) | 12 weeks
  Self-administered questionnaire measures the degree of reorganization (resolution) of internal conflict. Scores range from 0 to 110, with higher scores indicating higher level of internal conflict resolution.
Outcome Rating Scale | 12 weeks
  Self-administered visual analogue scale, measure of wellbeing. Scores range from 0 to 40, with higher scores indicating higher level of wellbeing.

IPD SHARING:
Plan to Share IPD: No